CLINICAL TRIAL: NCT00005041
Title: A Phase II Study to Determine the Antitumor Activity of Farnesyltransferase Inhibitor R115777 in Subjects With Relapsed Small Cell Lung Cancer
Brief Title: R115777 in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067632; NYU-9861; JRF-R115777-USA-8B; NCI-G00-1714
Record Dates: First submitted 2000-04-06; First posted 2004-06-18 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2000-11

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of R115777 in treating patients who have relapsed small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate (complete or partial) and duration of response of patients with small cell lung cancer who have had at least a partial response to one prior chemotherapy regimen for at least 3 months when treated with R115777. II. Determine the time to disease progression, survival, and quality of life in this patient population treated with this drug. III. Assess the safety of R115777 in this patient population. IV. Assess the presence of ras mutations in relapsed patients with available paraffin blocks.

OUTLINE: This is a multicenter study. Patients receive oral R115777 every 12 hours for 14 consecutive days followed by 7 days of rest. Treatment continues in the absence of unacceptable toxicity or disease progression. Quality of life is assessed at baseline, on day 15 of each course, and at the end of the study.

PROJECTED ACCRUAL: A total of 27-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed small cell lung cancer for which no potentially curative therapy exists Confirmation at relapse required only if sole relapse site is within previous radiation port No mixed histology Bidimensionally measurable disease by CT scan At least 1 measurable lesion at least 2 cm At least a partial response to front line chemotherapy Single regimen or alternating regimen allowed No initial course exceeding 8 courses or lasting more than 6 months No uncontrolled, untreated brain metastases No extensive liver metastases such that greater than 50% of liver parenchyma is replaced with metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if documented liver metastases) Renal: Creatinine less than 2.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study Adequate unassisted oral or adequate enteral intake to maintain reasonable state of nutrition No other concurrent medical condition that would preclude study therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow transplantation No concurrent immunotherapy No concurrent myeloid colony stimulating factors (e.g., filgrastim (G-CSF), sargramostim (GM-CSF), interleukin-11) Chemotherapy: See Disease Characteristics At least 3 months since prior chemotherapy measured from day 1 of last course of front line therapy No prior high dose chemotherapy with marrow or stem cell rescue No more than 1 prior chemotherapy regimen No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: At least 2 weeks since prior radiotherapy No prior extensive radiotherapy (greater than 25% of bone marrow) No concurrent radiotherapy except for patients who are responding and develop brain metastases Surgery: Not specified Other: At least 30 days since prior investigational drugs No concurrent participation in another investigational trial No other concurrent experimental agents No other concurrent anticancer therapy No prophylactic oral or IV antibiotics for neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Chachoua, MD, Study Chair — NYU Langone Health
Locations (1):
- Kaplan Cancer Center, New York, New York, United States